CLINICAL TRIAL: NCT05693285
Title: Preterm Birth and Biomarkers for Cardiovascular Disease
Acronym: BIO-PRETERM
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: UU
Record Dates: First submitted 2022-12-12; First posted 2023-01-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Preterm Birth; Cardiovascular Diseases
MeSH Terms: conditions — Premature Birth; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collected at two time points, in pregnancy and at follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm birth: Women with spontaneous preterm birth in first pregnancy
  Interventions: Other: No intervention
- Controls: Matched controls with spontaneous delivery in normal time in first pregnancy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Preterm birth is associated with maternal increased risk of cardiovascular disease later in life. In an observational case- control study, investigators want to evaluate whether women with preterm birth have increased levels of biomarkers for cardiovascular disease, to reveal potential pathophysiological mechanisms in common.

DETAILED DESCRIPTION:
Women with spontaneous preterm birth in first pregnancy and a group of matched controls with spontaneous birth in normal time where invited to participate in the study. Participants were identified from the Biobank of Pregnant Women in Uppsala. Levels of cardiovascular biomarkers will be analyzed in plasma samples from the pregnancy and at a follow-up visit where investigators also collect information about other cardiovascular risk factors and lipid status.

ELIGIBILITY:
Inclusion Criteria:

* Women identified as cases or controls

Exclusion Criteria:

* System inflammatory disease
* Smoking at the time of the pregnancy

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women were identified in the Uppsala Biobank of pregnant women at their first pregnancy. Investigators invited women identified as cases or controls to participate by one blood sample and a visit collecting information about cardiovascular risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Levels of Factor XII in plasma in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of Factor XII in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of complement C5 in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of complement C5 in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of apolipoprotein M in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of apolipoprotein M in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of fibrinogen in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of fibrinogen in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of plasma kallikrein in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of plasma kallikrein in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of vitamin D binding protein in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of vitamin D binding protein in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of cadherin -5 in women with preterm birth in compared to a control group with delivery in normal time. | spring 2023
  Levels of cadherin -5 in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.
Levels of growth/differentiation Factor-15 (GDF-15) in women with preterm birth in compared to a control group with delivery in normal time. preterm birth compared to a control group with delivery in normal time. | spring 2023
  Levels of growth/differentiation Factor-15 (GDF-15) in plasma will be analyzed at two times, both in the actual pregnancy and at a follow-up visit where information about cardiovascular risk factors and lipid status is collected.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Christersson, Principal Investigator — Uppsala University
Locations (1):
- Department of Medical Sciences, Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cederlof ET, Lager S, Larsson A, Sundstrom Poromaa I, Lindahl B, Wikstrom AK, Christersson C. Biomarkers associated with cardiovascular disease in women with spontaneous preterm birth: A case-control study. Acta Obstet Gynecol Scand. 2024 May;103(5):970-979. doi: 10.1111/aogs.14813. Epub 2024 Feb 20. PMID 38379394